CLINICAL TRIAL: NCT00662597
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled Multi-Center Study of ASA404 in Combination With Paclitaxel and Carboplatin as First-Line Treatment for Locally Advanced or Metastatic (Stage IIIb/IV) Non-Small Cell Lung Cancer (NSCLC)
Brief Title: ASA404 or Placebo in Combination With Paclitaxel and Carboplatin as First-Line Treatment for Stage IIIb/IV Non-Small Cell Lung Cancer
Acronym: ATRACT-1
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CASA404A2301
Record Dates: First submitted 2008-04-17; First posted 2008-04-21 (Estimated); Last update posted 2020-12-24 (Actual); Status verified 2012-05

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Tumor vascular disrupting agent; VDA; ASA404; non-small cell lung cancer; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — vadimezan; Carboplatin; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- ASA404 (Experimental)
  Interventions: Drug: ASA404; Drug: carboplatin; Drug: Paclitaxel
- ASA40 Placebo (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: ASA404
  Arms: ASA404
Drug: Placebo
  Arms: ASA40 Placebo
Drug: carboplatin
Drug: Paclitaxel

SUMMARY:
The purpose of this study is to determine if adding ASA404 to standard chemotherapy makes the cancer treatment more effective in patients with advanced lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed non-small cell carcinoma of the lung. (Histological or cytological specimens must be collected via surgical biopsy, brushing, washing or core needle aspiration of a defined lesion. Sputum cytology is not acceptable.)
2. Newly diagnosed Stage IIIb disease (malignant pleural effusion or pericardial effusion that have been confirmed cytologically) or Stage IV disease
3. No prior systemic antineoplastic treatment for Stage IIIb/IV non-small cell carcinoma of the lung (Prior neoadjuvant or adjuvant chemotherapy for earlier stage I/II NSCLC is allowed if 12 months or more prior to Baseline visit.)
4. Age ≥ 18 years old
5. WHO Performance Status of 0-1
6. Measurable or non-measurable disease per RECIST criteria (Post-text supplement 1)
7. Lab values within the range, as defined below, within 2 weeks of randomization:

   * Absolute neutrophils count (ANC) > 2.0 x 109/L
   * Platelets ≥ 100 x109/L
   * Hemoglobin ≥ 10 g/dL
   * Serum creatinine ≤ 1.5 x ULN (≤ 120 micro mol/L)
   * Serum bilirubin ≤ 1.5 x ULN (≤ 25 micro mol/L)
   * Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 x ULN (≤ 5 x ULN if liver metastases)
   * International Normalized Ratio (INR) or Prothrombin Time (PT) ≤ 1.5 x IULN (Sections 6.9.1 and 7.3.4.2)
   * Electrolyte values (potassium, calcium, magnesium) within > 1 x LLN and < 1 x ULN. Patients with corrected electrolyte values are eligible. See Sections 6.8.1 and 7.3.4.3.
   * Females of child-bearing potential must have negative serum pregnancy test (confirmation of negative urine pregnancy test within 72 hours prior to initial dosing).
8. Life expectancy ≥ 12 weeks
9. Written informed consent obtained according to local guidelines

Exclusion Criteria:

1. Patients having CNS metastases (Patients having any clinical signs of CNS metastases must have a CT or MRI of the brain performed to rule out CNS metastases in order to be eligible for study participation. Patients who have had brain metastases surgically removed or irradiated with no residual disease confirmed by imaging are allowed.).
2. Patients with a history of another primary malignancy ≤ 5 years, with the exception of non-melanoma skin cancer or cervical cancer in situ.
3. Radiotherapy ≤ 2 weeks prior to randomization. Patients must have recovered from all radiotherapy-related toxicities.
4. Major surgery ≤ 4 weeks prior to randomization or minor surgery ≤ 2 weeks prior to randomization.(Major surgery is defined by the use of general anesthesia however, endoscopic examinations with diagnostic intent are not considered major surgery. Insertion of a vascular access device is exempt from this exclusion criteria. Patients must have recovered from all surgery-related complications.
5. Concurrent use of other investigational agents and patients who have received investigational agents ≤ 4 weeks prior to randomization
6. Prior exposure to Tumor-VDAs or other vascular targeting agents (anti-VEGF, anti-VEGF receptor agents, anti-EGFR agents [bevacizumab, cetuximab, etc.])
7. Pleural effusion that causes ≥ CTC grade 2 dyspnea
8. Patients with systolic BP > 160 mm Hg and/or diastolic BP >90 mm Hg
9. Patients with recent hemoptysis associated with NSCLC (> 1 teaspoon in a single episode within 4 weeks)
10. Patients with any one of the following:

    * Patients with long QT syndrome
    * Patients with a Baseline 12-lead ECG QTc of > 450 msec per central evaluation
    * Congestive heart failure (NY Heart Association class III or IV)
    * Patients with a myocardial infarction within 12 months of study entry
    * Unstable or poorly controlled angina pectoris, including Prinzmetal variant angina pectoris
    * History of labile hypertension or poor compliance with anti-hypertensive regimen
    * History of a sustained ventricular tachycardia
    * Any history of ventricular fibrillation or Torsades de Pointes
    * Right bundle branch block and left anterior hemiblock (bifasicular block)
    * Bradycardia defined as heart rate < 50 beats per minute
11. Concomitant use of drugs with a risk of causing Torsades de Pointes (See Table 6-3)
12. Known allergy or hypersensitivity to platinum-containing drugs, taxanes, other drugs formulated in Cremophor EL (polyoxyethylated castor oil) or any known excipients of these drugs.
13. Peripheral sensory neuropathy with functional impairment (CTC grade 2 neuropathy, regardless of causality)
14. Pregnant or breast feeding females

    • Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test (> 5 mIU/ml)
15. Women of child bearing potential or sexually active males, unwilling or unable to use the required highly effective method(s) of contraception for both sexes while receiving treatment and for at least 6 months after the discontinuation of study treatment. (Adequate forms of contraception include IUD, oral or depot contraceptive or the barrier method plus spermicide.)

    • Oral, implantable, or injectable contraceptives may be affected by cytochrome P450 interactions while taking paclitaxel and therefore are not considered effective contraceptive methods for this study when used as a single agent. Therefore, it is highly recommended that a concomitant barrier method be used with oral, implantable, or injectable contraceptives. The investigator shall counsel the patient accordingly. Women of childbearing potential must have a negative pregnancy test (serum or urine) 72 hours prior to administration of study treatment. For a list of substrates of human liver microsomal P450 enzymes, visit website (http://medicine.iupui.edu/flockhart/)
16. Concurrent severe and/or uncontrolled medical disease (i.e. uncontrolled diabetes, chronic renal disease, chronic liver disease, confirmed diagnosis of HIV infection or active uncontrolled infection).
17. Significant neurologic or psychiatric disorder which could compromise participation in the study Patient unwilling or unable to comply with the protocol

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1285 (Actual)
Dates: Start 2008-04; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Overall survival rate | Patients will be followed every six weeks for survival following treatment completion, discontinuation, or documented disease progression until either death or the data cut off date.

SECONDARY OUTCOMES:
Overall survival of patients with squamous and non-squamous NSCLC | Patients will be followed every six weeks for survival following treatment completion, discontinuation, or documented disease progression until either death or the data cut off date.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (248):
- United States (100):
  - University of South Alabama/Mitchell Cancer Institute, Mobile, Alabama
  - Arizona Oncology Associates, Tucson, Arizona
  - University of Arizona Cancer Center, Tucson, Arizona
  - Highlands Oncology Group, Bentonville, Arkansas
  - Genesis Cancer Center, Hot Springs, Arkansas
  - Alta Bates Summit Medical Center, Berkeley, California
  - Pacific Oncology and Hematology Association, Encinitas, California
  - Cancer Care Associates, Fresno, California
  - Ronald Yanagihara - Private Practice, Gilroy, California
  - California Cancer Care, Greenbrae, California
  - Moores UCSD Cancer Center, La Jolla, California
  - Loma Linda University Cancer Center, Loma Linda, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - University of California Irvine Comprhensive Center, Orange, California
  - Loma Linda Oncology Medical Group, Inc., Redlands, California
  - UC Davis Comprehensive Cancer Center, Sacramento, California
  - California Pacific Medical Research Institute, San Francisco, California
  - Redwood Regional Cancer Center, Santa Rosa, California
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Palm Beach Institute of Hematology & Oncology, Boynton Beach, Florida
  - Florida Cancer Specialists, Bradenton, Florida
  - Cancer Centers of Central Florida, PA, Leesburg, Florida
  - Advanced Medical Specialties (ACORN), Miami, Florida
  - Northwest Georgia Oncology Centers, Marietta, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Kootenai Cancer Center (ACORN), Coeur d'Alene, Idaho
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - Illinois Oncology/Warren Billhartz Cancer Ctr., Maryville, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Hematology/Oncology of North Shore, Skokie, Illinois
  - Loyola Cancer Care & Research Ctr. at Central Dupage Hospital, Winfield, Illinois
  - Ft. Wayne Oncology and Hematology, Fort Wayne, Indiana
  - Siouxland Hematology-Oncology Assoc., LLC, Sioux City, Iowa
  - Kansas City Cancer Center, Southwest, Overland Park, Kansas
  - University of Louisville - James Graham Brown Cancer Center, Louisville, Kentucky
  - Hematology Oncology Specialists, Metairie, Louisiana
  - Louisiana State University Health Sciences Center - Feist-Weiller Cancer Center, Shreveport, Louisiana
  - St. Agnes Cancer Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore - The Alvin & Lois Lapidus Cancer Institute, Baltimore, Maryland
  - The Harry and Jeanette Weinberg Cancer Institute at Franklin Square/MedStar Health, Baltimore, Maryland
  - Peninsula Regional Oncology and Hematology, Salisbury, Maryland
  - Boston VA Healthcare System, Boston, Massachusetts
  - Fallon Clinic, Worcester, Massachusetts
  - Breslin Cancer Center, Lansing, Michigan
  - Osteopathic Medical Oncology and Hematology PC, Woodhaven, Michigan
  - St. Luke's Hospital - St Luke's Cancer Center, Duluth, Minnesota
  - Kansas City Veterans Affair Medical Center, Kansas City, Missouri
  - St. Louis University Cancer Center, St Louis, Missouri
  - Center for Cancer Care and Research (US Oncology), St Louis, Missouri
  - St. John's Mercy Medical Center, St Louis, Missouri
  - St. Louis Cancer and Breast Institute, St Louis, Missouri
  - Billings Clinic, Billings, Montana
  - Sletten Cancer Institute, Great Falls, Montana
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Arena Oncology Associates, Lake Success, New York
  - New York Oncology Hematology, Latham, New York
  - Hematology Oncology Associates of Rockland, Nyack, New York
  - Rochester General Hospital - Lipson Cancer Center, Rochester, New York
  - Syracuse VA Medical Center, Syracuse, New York
  - Eastchester Center for Cancer Care, The Bronx, New York
  - Alamance Regional Medical Center-Cancer Ctr., Burlington, North Carolina
  - Carolina Cancer Mgmt/Cape Fear Valley Health System/Med Onc, Fayetteville, North Carolina
  - Akron City Hospital, Akron, Ohio
  - Oncology Hematology Care Research, Cincinnati, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Medical Oncology Hematology Associates, Inc. - Dayton Clinical Oncology Program, Dayton, Ohio
  - Medical Oncology Hematology Associates, Inc., Dayton, Ohio
  - Cleo Craig Memorial Cancer Ctr. & Research Clinic, Lawton, Oklahoma
  - University of Oklahoma Health Science Center, Oklahoma City, Oklahoma
  - Kaiser Permanente, Northwest Region, Portland, Oregon
  - Allegheny General Hospital/Allegheny Cancer Center, Pittsburgh, Pennsylvania
  - South Carolina Oncology Associate, Columbia, South Carolina
  - Lowcountry Hematology & Oncology PA, Mt. Pleasant, South Carolina
  - Chattanooga Oncology Hematology Associates, Chattanooga, Tennessee
  - The West Clinic, Memphis, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
  - Texas Oncology Cancer Center of the High Plains, Amarillo, Texas
  - Arlington Cancer Center, Arlington, Texas
  - Patient's Comprehensive Cancer Center, Carrollton, Texas
  - South Texas Cancer Institute, Corpus Christi, Texas
  - Cancer Care Centers of South Texas, Dallas, Texas
  - Texas Oncology at Presbyterian Hospital, Dallas, Texas
  - University of Texas Southwestern Medical Center/Simmons Comprehensive Cancer Center, Dallas, Texas
  - Texas Oncology at Garland, Garland, Texas
  - HOPE Oncology, Richardson, Texas
  - Tyler Cancer Center, Tyler, Texas
  - UT Health Center, Tyler, Texas
  - Deke Slayton Cancer Center, Webster, Texas
  - Texoma Cancer Center, Wichita Falls, Texas
  - Northern Utah Associates, Ogden, Utah
  - Danville Hematology & Oncology, Danville, Virginia
  - Medical Oncology & Hematology Associates of Northern Virginia, Fairfax, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - Highline Medical Oncology, Burien, Washington
  - Providence Everett Medical Center/Providence regional Cancer Partnership, Everett, Washington
  - Northwest Cancer Specialists, Vancouver, Washington
  - University of Wisconsin, Madison, Wisconsin
  - Medical Consultants, Milwaukee, Wisconsin
  - Medical College of Wisconsin/Division of Neoplastic & Related Disorders, Milwaukee, Wisconsin
- Argentina (6):
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, Capital Federal
  - Novartis Investigative Site, Córdoba
  - Novartis Investigative Site, La Plata
  - Novartis Investigative Site, Mendoza
  - Novartis Investigative Site, Rosario
- Australia (3):
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Herston
  - Novartis Investigative Site, South Brisbane
- Belgium (3):
  - Novartis Investigative Site, Duffel
  - Novartis Investigative Site, Jette
  - Novartis Investigative Site, Liège
- Brazil (8):
  - Novartis Investigative Site, Barretos
  - Novartis Investigative Site, Belo Horizonte
  - Novartis Investigative Site, Goiânia
  - Novartis Investigative Site, Jaù
  - Novartis Investigative Site, Jaú
  - Novartis Investigative Site, Porto Alegre
  - Novartis Investigative Site, Santo André
  - Novartis Investigative Site, São Paulo
- Canada (10):
  - Novartis Investigative Site, Calgary
  - Novartis Investigative Site, Greenfield Park
  - Novartis Investigative Site, Kitchener
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Moncton
  - Novartis Investigative Site, Montreal
  - Novartis Investigative Site, Rimouski
  - Novartis Investigative Site, Sainte-Foy
  - Novartis Investigative Site, Sherbrooke
  - Novartis Investigative Site, Sult Ste-Marie
- China (5):
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Guangzhou
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Wuhan
  - Novartis Investigative Site, Xi'an
- Czechia (3):
  - Novartis Investigative Site, Brno
  - Novartis Investigative Site, Ostrava Poruba
  - Novartis Investigative Site, Prague
- France (12):
  - Novartis Investigative Site, Bobigny
  - Novartis Investigative Site, Boujan-sur-Libron
  - Novartis Investigative Site, Clamart
  - Novartis Investigative Site, Le Mans
  - Novartis Investigative Site, Limoges
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Saint-Herblain
  - Novartis Investigative Site, Toulon Armées
  - Novartis Investigative Site, Tours
- Germany (16):
  - Novartis Investigative Site, Aschaffenburg
  - Novartis Investigative Site, Bad Berka
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Donaustauf
  - Novartis Investigative Site, Ebensberg
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Gerlingen
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Grosshandsdorf
  - Novartis Investigative Site, Heidenheim
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Merseburg
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Nuremberg
- Greece (3):
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Heraklion Crete
  - Novartis Investigative Site, Thessaloniki
- Novartis Investigative Site, Hong Kong, Hong Kong
- Hungary (3):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Deszk
  - Novartis Investigative Site, Mátraháza
- Israel (5):
  - Novartis Investigative Site, Kfar Saba
  - Novartis Investigative Site, Rehovot
  - Novartis Investigative Site, Tel Aviv
  - Novartis Investigative Site, Tel Litwinsky
  - Novartis Investigative Site, Zrifin
- Italy (8):
  - Novartis Investigative Site, Avellino
  - Novartis Investigative Site, Milan
  - Novartis Investigative Site, Modena
  - Novartis Investigative Site, Napoli
  - Novartis Investigative Site, Orbassano
  - Novartis Investigative Site, Parma
  - Novartis Investigative Site, Perugia
  - Novartis Investigative Site, Roma
- Japan (19):
  - Novartis Investigative Site, Akashi
  - Novartis Investigative Site, Fukuoka
  - Novartis Investigative Site, Habikino
  - Novartis Investigative Site, Hiroshima
  - Novartis Investigative Site, Kashiwa
  - Novartis Investigative Site, Kobe
  - Novartis Investigative Site, Kōtō City
  - Novartis Investigative Site, Kumamoto
  - Novartis Investigative Site, Kurashiki
  - Novartis Investigative Site, Matsuyama
  - Novartis Investigative Site, Nagoya
  - Novartis Investigative Site, Niigata
  - Novartis Investigative Site, Okayama
  - Novartis Investigative Site, Osaka
  - Novartis Investigative Site, Ōsaka-sayama
  - Novartis Investigative Site, Sapporo
  - Novartis Investigative Site, Sendai
  - Novartis Investigative Site, Ube
  - Novartis Investigative Site, Yokohama
- Netherlands (6):
  - Novartis Investigative Site, 's-Hertogenbosch
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Breda
  - Novartis Investigative Site, Eindhoven
  - Novartis Investigative Site, Harderwijk
  - Novartis Investigative Site, Zwolle
- New Zealand (4):
  - Novartis Investigative Site, Auckland
  - Novartis Investigative Site, Christchurch
  - Novartis Investigative Site, Hamilton
  - Novartis Investigative Site, Wellington
- Poland (4):
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Lublin
  - Novartis Investigative Site, Otwock
  - Novartis Investigative Site, Poznan
- Novartis Investigative Site, Singapore, Singapore
- South Korea (3):
  - Novartis Investigative Site, Seoul
  - Novartis Investigative Site, Seungnam
  - Novartis Investigative Site, Suwon
- Spain (9):
  - Novartis Investigative Site, Barakaldo
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Córdoba
  - Novartis Investigative Site, Granada
  - Novartis Investigative Site, Jaén
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Pontevedra
  - Novartis Investigative Site, Seville
  - Novartis Investigative Site, Zaragoza
- Novartis Investigative Site, Umeå, Sweden
- Taiwan (5):
  - Novartis Investigative Site, Kaoshiung
  - Novartis Investigative Site, Lin-Ko
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Tainan
  - Novartis Investigative Site, Taipei
- Turkey (Türkiye) (4):
  - Novartis Investigative Site, Altunizade
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Izmir
- United Kingdom (6):
  - Novartis Investigative Site, Aberdeen
  - Novartis Investigative Site, Cambridge
  - Novartis Investigative Site, Leicester
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Sutton

REFERENCES:
- See also: Results for CASA404A2301 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=4609